CLINICAL TRIAL: NCT00521157
Title: Naltrexone Naltrexone Implants as an Aid in Preventing Relapse Following Inpatient Treatment for Opioid Addiction - a Randomised Study
Brief Title: Naltrexone Implants as an Aid in Preventing Relapse Following Inpatient Treatment for Opioid Addiction
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Oslo (Other)
Responsible Party: Helge Waal, MD, Professor, Head of Center for Addiction Research, University of Oslo, Institute of Psychiatry, University of Oslo
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 11899 revised
Record Dates: First submitted 2007-08-24; First posted 2007-08-27 (Estimated); Last update posted 2009-05-05 (Estimated); Status verified 2009-05

CONDITIONS: Opiate Dependence
Keywords: Substance abuse; Opiate dependency; Treatment; Relapse prevention
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- intervention (Experimental): Experimental group randomised after abstinence oriented treatment
  Interventions: Drug: Go Medical Naltrexone implants
- 2 (No Intervention): waiting list control

INTERVENTIONS:
Drug: Go Medical Naltrexone implants — Naltrexone implants 3.2 g (double of 1,6 g)
  Other Names: Go Medical naltrexone implant
  Arms: intervention

SUMMARY:
The purpose of this clinical trial is to study the efficacy and safety of naltrexone implants as relapse prevention for patients that are completing treatment for opiate addiction in inpatient (or similarly controlled) settings. Participants volunteer for the study before being released from inpatient treatment, and are randomized to a naltrexone implant group or a waiting-list control for the duration of the first six months following completion of inpatient treatment. Both groups are free to receive treatment as usual (TAU) from the Norwegian healthcare system. After six months, both groups will be offered to have naltrexone implanted for the remaining six months of the study.

The hypotheses are that quality of life, depression, opioid use, will be significantly better in the naltrexone group compared to the non at 6-month follow-up. For the last six months of the trial, the investigators hypothesise that choice of naltrexone implant will mainly strengthen positive tendencies or reverse negative trends on the aforementioned variables.

The investigators also hypothesize that the implants can prevent death from opioid overdose up to 6 months after commenced treatment.

ELIGIBILITY:
Inclusion Criteria:

* soon to complete inpatient treatment for opioid addiction
* living in southern Norway

Exclusion Criteria:

* psychosis/major depression, currently not treated
* pregnancy
* liver enzymes: ASAT or ALAT > threefold above upper boundary
* maintenance treatment with methadone or buprenorphine

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2006-01; Primary Completion 2008-06 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Drug use at 6 (12) months by self report and hair analysis | 6 and 12 months
Days in work or education | 6 and 12 months
Number of drug-free friends at 6 (12) months by self report | 6 and 12 months

SECONDARY OUTCOMES:
Depression at 6 (12) months by BDI and Hopkins SCL-25 | 6 and 12 months
Quality of life at 6 (12) months by EuropASI | 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Helge Waal, Professor, Study Director — Unit for addiction medicine, Institute of psychiatry, University of Oslo; Helge Waal, MD, Study Director — Norwegian Medical Association
Locations (1):
- Unit for Addiction Medicine, University of Oslo, Oslo, Norway

REFERENCES:
- [Derived] Kornor H, Lobmaier PPK, Kunoe N. Sustained-release naltrexone for opioid dependence. Cochrane Database Syst Rev. 2025 May 9;5(5):CD006140. doi: 10.1002/14651858.CD006140.pub3. PMID 40342086
- [Derived] Kunoe N, Lobmaier P, Vederhus JK, Hjerkinn B, Gossop M, Hegstad S, Kristensen O, Waal H. Challenges to antagonist blockade during sustained-release naltrexone treatment. Addiction. 2010 Sep;105(9):1633-9. doi: 10.1111/j.1360-0443.2010.03031.x. PMID 20707781